CLINICAL TRIAL: NCT02129023
Title: The Impact of Exergame on User Health: A Randomized Controlled Trial
Brief Title: The Impact of Exergame on User Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung University (Other)
Collaborators: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Ching-I Teng, Professor, Chang Gung University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: CMRPD3D0021
Record Dates: First submitted 2014-04-15; First posted 2014-05-01 (Estimated); Last update posted 2019-02-05 (Actual); Status verified 2019-02

CONDITIONS: Impact of Exergame Use on User Health
Keywords: Exergame; user health; exercise
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- exergame (Experimental): Participants were asked to use exergame (Xbox 360) half hour for three times per week in the 12-week study period.
  Interventions: Device: Xbox 360
- control (No Intervention): Participants were not asked to use exergames.

INTERVENTIONS:
Device: Xbox 360 — For each participant in the experimental arm, two Xbox 360 exercise items were randomly selected from the nine items, which are related to user health. Each participant takes the two exercise items in turn.
  Arms: exergame

SUMMARY:
The purpose of this study is to examine whether exergame use can improve user health, in terms of physical fitness, self-rated mental health and physical health, and favorable attitude, strong intention, and actual behavior of future exercise. Moreover, this study also examines whether past exercise moderates the impact of exergame use on user health.

DETAILED DESCRIPTION:
The main hypotheses are:

H1: Compared with the control group participants (who do not use exergame) the experimental group participants (who use exergame) have better change in physical fitness. The difference between these two groups in the amount of change is negatively related to past exercise.

H2: Compared with the control group participants (who do not use exergame) the experimental group participants (who use exergame) have better change in (a) mental health and (b) physical health after the intervention. The difference between these two groups in the amount of change is negatively related to past exercise.

H3: Compared with the control group participants (who do not use exergame) the experimental group participants (who use exergame) have better change in (a) attitude, (b) intention and (c) behavior of doing another exercise in the future. The difference between these two groups in the amount of change is negatively related to past exercise.

ELIGIBILITY:
Inclusion Criteria:

* junior and senior undergraduate student
* senior graduate student

Exclusion Criteria:

* asthma
* high myopia
* anemia
* vertigo
* cardiopathy
* hypertension
* unstable of intracranial pressure and blood pressure
* cardiac arrhythmia
* heart failure
* angor pectoris
* injury of vertebra
* ankylosing spondylitis
* hereditary cardiac arrhythmia
* musculoskeletal system injury
* glaucoma
* psychiatric disorders

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2014-01 (Actual); Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Change in physical fitness | The beginning and the end of expected average of 12 weeks
  Physical fitness was assessed twice by Chang Gung Memorial Hospital, including body composition, cardio-pulmonary function, muscular strength, muscular endurance, explosive force, flexibility, agility, sense of balance, and cardiorespiratory endurance.

SECONDARY OUTCOMES:
Change in mental and physical health (12 weeks) | The beginning and the end of expected average of 12 weeks
  Self-rated mental and physical health, using the SF-36 scale.
Change in attitude of future exercise (12 weeks) | The beginning and the end of expected average of 12 weeks
  Self-reported questionnaires assessing users' attitude toward future exercise between an expected average of 12 weeks since randomization.
Change in intention of future exercise (12 weeks) | The beginning and the end of expected average of 12 weeks
  Self-reported questionnaires assessing users' intention to do exercise in the future between an expected average of 12 weeks since randomization.
Change in behavior of future exercise (12 weeks) | The beginning and the end of expected average of 12 weeks
  Self-reported questionnaires assessing users' actual exercise behavior between an expected average of 12 weeks since randomization.
Change in mental and physical health (8 weeks) | The beginning and the end of expected average of 8 weeks
  Self-rated mental and physical health, using the SF-36 scale.
Change in attitude of future exercise (8 weeks) | The beginning and the end of expected average of 8 weeks
  Self-reported questionnaires assessing users' attitude toward future exercise between an expected average of 8 weeks since randomization.
Change in intention of future exercise (8 weeks) | The beginning and the end of expected average of 8 weeks
  Self-reported questionnaires assessing users' intention to do exercise in the future between an expected average of 8 weeks since randomization.
Change in behavior of future exercise (8 weeks) | The beginning and the end of expected average of 8 weeks
  Self-reported questionnaires assessing users' actual exercise behavior between an expected average of 8 weeks since randomization.
Change in mental and physical health (4 weeks) | The beginning and the end of expected average of 4 weeks
  Self-rated mental and physical health, using the SF-36 scale.
Change in attitude of future exercise (4 weeks) | The beginning and the end of expected average of 4 weeks
  Self-reported questionnaires assessing users' attitude toward future exercise between an expected average of 4 weeks since randomization.
Change in intention of future exercise (4 weeks) | The beginning and the end of expected average of 4 weeks
  Self-reported questionnaires assessing users' intention to do exercise in the future between an expected average of 4 weeks since randomization.
Change in behavior of future exercise (4 weeks) | The beginning and the end of expected average of 4 weeks
  Self-reported questionnaires assessing users' actual exercise behavior between an expected average of 4 weeks since randomization.

OTHER OUTCOMES:
Perceived Challenge (beginning) | Beginning of the participation in this study
  Evaluated using scales measuing perceived challenge
Perceived Achievement (beginning) | Beginning of the participation in this study
  Evaluated using scales measuing perceived achievement
Continuance Intention (beginning) | Beginning of the participation in this study
  Evaluated using scales measuing intention to continue to use the exergame
Perceived Challenge (after 4 weeks) | After 4 weeks of the participation in this study
  Evaluated using scales measuing perceived challenge
Perceived Achievement (after 4 weeks) | After 4 weeks of the participation in this study
  Evaluated using scales measuing perceived achievement
Continuance Intention (after 4 weeks) | After 4 weeks of the participation in this study
  Evaluated using scales measuing intention to continue to use the exergame
Perceived Challenge (after 8 weeks) | After 8 weeks of the participation in this study
  Evaluated using scales measuing perceived challenge
Perceived Achievement (after 8 weeks) | After 8 weeks of the participation in this study
  Evaluated using scales measuing perceived achievement
Continuance Intention (after 8 weeks) | After 8 weeks of the participation in this study
  Evaluated using scales measuing intention to continue to use the exergame
Perceived Challenge (after 12 weeks) | After 12 weeks of the participation in this study
  Evaluated using scales measuing perceived challenge
Perceived Achievement (after 12 weeks) | After 12 weeks of the participation in this study
  Evaluated using scales measuing perceived achievement
Continuance Intention (after 12 weeks) | After 12 weeks of the participation in this study
  Evaluated using scales measuing intention to continue to use the exergame

CONTACTS AND LOCATIONS:
Overall Officials: Ching-I Teng, PhD, Principal Investigator — Chang Gung University
Locations (1):
- Chang Gung University, Taoyuan District, Taiwan